CLINICAL TRIAL: NCT05851261
Title: Phase I Clinical Study to Evaluate the Safety, Tolerance, Pharmacokinetics Characteristics of Single and Multiple Administration of Oral PA3670 Tablets in Chinese Healthy Subjects and the Effect of Food on Pharmacokinetics
Brief Title: Study to Evaluate the Safety, Tolerance, Pharmacokinetics Characteristics of PA3670 Tablets in Chinese Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Zhejiang Palo Alto Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PA3670-101
Record Dates: First submitted 2023-02-08; First posted 2023-05-09 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Chronic HBV Infection

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- PA3670 5 mg (Placebo Comparator): Ten subjects will be randomly assigned in a ratio of 4:1 to receive 5 mg of PA3670 tablets or PA3670 placebo tablets. They will be administered a single dose and observed for four days.
  Interventions: Drug: PA3670
- PA3670 15 mg (Placebo Comparator): Ten subjects will be randomly assigned in a ratio of 4:1 to receive 15 mg of PA3670 tablets or PA3670 placebo tablets. They will be administered a single dose and observed for four days.
  Interventions: Drug: PA3670
- PA3670 30 mg (Placebo Comparator): Ten subjects will be randomly assigned in a ratio of 4:1 to receive 30 mg of PA3670 tablets or PA3670 placebo tablets. They will be administered a single dose and observed for four days.
  Interventions: Drug: PA3670
- PA3670 15 mg for 9days (Placebo Comparator): Ten subjects will be randomly assigned at a 4: 1 ratio to receive either 15mg of PA3670 tablets or PA3670 placebo tablets, once daily for 9 days.
  Interventions: Drug: PA3670
- PA3670 15mg before and after meals (Other): Ten subjects will be administered 15mg PA3670 after overnight fasting for 10 hours in the first cycle, and then will be administered 10mg PA3670 within 30 minutes after high-fat meal in the second cycle. They will receive a single dose in each cycle and will be observed for four days. The cleaning period between the two cycles is more than 7 days.
  Interventions: Drug: PA3670
- PA3670 15mg after and before meals (Other): Ten subjects will be administered 15mg PA3670 within 30 minutes after the high-fat meal in the first cycle, and then will be administered 10mg PA3670 after overnight fasting 10 hours in the second cycle. They will receive a single dose in each cycle and will be observed for four days. The cleaning period between the two cycles is more than 7 days.
  Interventions: Drug: PA3670

INTERVENTIONS:
Drug: PA3670 — Placebo as control

SUMMARY:
The primary objectives of this study are to evaluate the safety and tolerance of single and multiple oral administration of PA3670 tablets in Chinese adult healthy subjects and the effect of food on pharmacokinetics of PA3670 tablets in Chinese adult healthy subjects.

DETAILED DESCRIPTION:
Stage I: Single dose, Single Ascending Dose (SAD) This is a randomized, double-blind, placebo-controlled, dose-escalation clinical trial.

The objective is to evaluate the safety, tolerability and pharmacokinetics characteristics of PA3670 tablets in Chinese healthy subjects. There are three dose groups of PA3670(5 mg、15 mg、30 mg) proposed to be tested sequentially in this study. A total of 30 healthy subjects are planned to be enrolled in this study and will be randomly assigned to the corresponding dose group in equal proportion, stratified by gender (male vs female). 10 subjects in each dose group are randomly assigned in a ratio of 4:1 to receive PA3670 tablets or placebo. All subjects will be dosed in a single dose, and the dose-related safety, tolerability and PK of PA3670 will be evaluated.

Stage Ⅱ: Multiple dose This is a randomized, double-blind, placebo-controlled, multiple dose clinical trial. A total of 10 subjects are planned to be enrolled in this study and will be randomly assigned in a ratio of 4:1 to receive 15mg PA3670 tablets or placebo. All subjects will be dosed for 9 consecutive days, and safety, tolerability and PK of PA3670 will be evaluated.

Stage Ⅲ: Study on the effect of food on Pharmacokinetics This is a randomized, open, two group crossover clinical trial. A total of 20 subjects are planned to be enrolled in this study, and will be randomly assigned to a dosing order (i.e. fasting administration followed by high-fat meal administration, or high-fat meal administration followed by fasting administration) in a ratio of 1:1. Subjects will be dosed 15 mg PA3670 tablets in a single dose, and the food-related PK of PA1010 will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* 1. Healthy male and female subjects aged from 18 to 65 (inclusive);
* 2. Male weight ≥ 50 kg, female weight ≥ 45 kg, and body mass index (BMI) between 19 and 28 kg/m2 (including the critical value);
* 3. Be able to complete the test according to the study protocol;
* 4. Voluntary participation and signing of informed consent.

Exclusion Criteria:

* 1. There are any medical conditions that the investigator thinks may increase the risk of the subject participating in the study (especially the history of esophageal or gastrointestinal ulcer), may interfere with drug absorption, distribution, metabolism or excretion, or may weaken the compliance of the study protocol;
* 2. Allergic to the study drug or any component of the study drug, or allergic (refers to allergic to 2 or more kinds of food, drugs or environmental substances);
* 3. The vital signs, physical examination, laboratory examination (blood routine test, blood biochemistry, urine routine test, blood coagulation function, etc.), chest X-ray examination, abdominal B-ultrasound (liver, gallbladder, pancreas, spleen, kidney), 12 lead ECG, etc. in the screening period were judged abnormal and had clinical significance;
* 4. Those who are positive for hepatitis B surface antigen, hepatitis C virus antibody, treponema pallidum antibody and HIV antibody;
* 5. Those who regularly drank alcohol within 3 months before screening, i.e., those who drank more than 14 units of alcohol every week (1 unit=360 mL of beer with 5% alcohol content, 45 mL of spirits with 40% alcohol content, or 150 mL of wine with 12% alcohol content), or those who had positive alcohol breath test in the baseline period or could not stop drinking alcohol during the study period;
* 6. Those who smoke ≥ 5 cigarettes a day within 3 months before screening, those who are positive for nicotine test in the baseline period, or those who cannot stop using any tobacco products during the test period;
* 7. Those who have a history of drug abuse and drug abuse in the past two years, or who are positive for urine screening of drug abuse at baseline (including morphine, methamphetamine, ketamine, benzodiazepine, cocaine, tetrahydrocannabinol acid);
* 8. Those who have used any drugs (prescription drugs, over-the-counter drugs, Chinese herbal medicine, vaccines) or health products within 4 weeks before screening and during screening;
* 9. Those who take any food or drink rich in caffeine and xanthine (coffee, tea, cola, chocolate, seafood, animal liver, etc.) within 48 hours before the first use of the study drug, or do not agree to stop eating the above diet during the test period;
* 10. Female subjects had unprotected sex in the past two weeks; Male subjects (or their partners) or female subjects who have fertility plans or donated sperm and eggs during the whole test period and within 3 months after administration, and who are unwilling to take one or more physical contraceptive measures or are breastfeeding during the test period;
* 11. Those who donate blood or lose a lot of blood (≥ 200 mL, except female physiological period) or use blood products or transfusions within 90 days before screening and during screening;
* 12. Those who participated in other clinical study within 90 days before screening or who participated in other clinical trials for less than 7 days;
* 13. Those who have undergone major surgery within 6 months before screening (judged by the researcher based on previous medical history data), suffered major trauma or planned to undergo surgery during the study period;
* 14. Difficulty in venous blood collection, or known history of needle and blood fainting;
* 15. Positive blood pregnancy test during screening period;
* 16. The investigator considers that there are other circumstances that are not suitable for participating in the test.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-04-13 (Actual); Primary Completion 2023-10-24 (Actual); Study Completion 2023-12-19 (Actual)

PRIMARY OUTCOMES:
Body temperature | Up to 72 hours after last dose
  Vital sign-body temperature
Systolic and diastolic blood pressure | Up to 72 hours after last dose
  Vital sign-Systolic and diastolic blood pressure
Pulse rate | Up to 72 hours after last dose
  Vital sign-Pulse rate
Breathing rate | Up to 72 hours after last dose
  Vital sign-Breathing rate
Number of subjects having abnormal hematology laboratory parameters | Up to 72 hours after last dose
  Absolute and relative number of subjects with values below, within or above the normal range will be assessed.
Number of subjects with abnormal clinical chemistry parameters | Up to 72 hours after last dose
  Absolute and relative number of subjects with values below, within or above the normal range will be assessed.
Number of subjects with abnormal values for urinalysis | Up to 72 hours after last dose
  Absolute and relative number of subjects with values below, within or above the normal range will be assessed.
Number of subjects with abnormal with blood coagulation function | Up to 72 hours after last dose
  Absolute and relative number of subjects with values below, within or above the normal range will be assessed.
ECG parameter-QTc interval | Up to 72 hours after last dose
  A 12-lead electrocardiogram (ECG) will be recorded using an ECG machine that automatically measures QTc interval
ECG parameter-PR interval | Up to 72 hours after last dose
  A 12-lead electrocardiogram (ECG) will be recorded using an ECG machine that automatically measures PR interval.
ECG parameter-QRS duration | Up to 72 hours after last dose
  A 12-lead electrocardiogram (ECG) will be recorded using an ECG machine that automatically measures QRS duration
Number of subjects experiencing adverse events (AEs) | 7 days or 15 days
  An adverse event (AE) is defined as any untoward medical occurrence in a clinical study subject administered a medicinal product which does not necessarily have a causal relationship with this treatment.

SECONDARY OUTCOMES:
Pharmacokinetics of PA3670-Cmax | 4 days or 12 days
  Blood samples will be collected serially, and the concentrations of PA3670 in plasma samples are determined by liquid chromatography/mass spectrometry/mass spectrometry (LC/MS/MS), followed by the calculation of pharmacokinetic parameter Maximum Observed Plasma Concentration (Cmax)
Pharmacokinetics of PA3670-Tmax | 4 days or 12 days
  Blood samples will be collected serially, and the concentrations of PA3670 in plasma samples are determined by liquid chromatography/mass spectrometry/mass spectrometry (LC/MS/MS), followed by the calculation of pharmacokinetic parameter Time to Reach Maximum Observed Plasma Concentration (Tmax)
Pharmacokinetics of single dose of PA3670-AUC | 4 days or 12 days
  Blood samples will be collected serially, and the concentrations of PA3670 in plasma samples are determined by liquid chromatography/mass spectrometry/mass spectrometry (LC/MS/MS), followed by the calculation of pharmacokinetic parameter Area Under the Plasma Concentration-Time Curve (AUC)

CONTACTS AND LOCATIONS:
Overall Officials: Hong Ren, MD, Principal Investigator — The Second Affiliated Hospital of Chongqing Medical University
Locations (1):
- The Second Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China